CLINICAL TRIAL: NCT03105063
Title: Evaluation of the AIIS Using Hip Ultrasound(AIISUS)
Acronym: AIISUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-17-RA-846-CTIL
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: AIS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- US GROUP (Experimental): All patients will first undergo ultrasound scan of the hip in attempt to recognize the AIIS, on the same day , the true morphology of the AIIS will be evaluated using 3d imaging
  Interventions: Diagnostic Test: ultrasound scan of the hip

INTERVENTIONS:
Diagnostic Test: ultrasound scan of the hip — validation of Ultrasound test as a tool for diagosing AIIS morphology

SUMMARY:
The anatomy of the acetabulum is well described in the past literature, yet the understanding of the clinical importance of the anatomical morphology of the AIIS has grown in recent years. Hetsroni et al. (2013) proposed a morphological classification of AIIS. In this classification, three types AIIS are identified based on the relationship between the distal extension of the acetabular rim and the AIIS. Unfortunately classifying the morphology of the AIIS using standard AP pelvis examination is misleading and requires additional imagery, a specific radiographic projection - false profile pelvis or 3d imaging techniques such as CT or MRI.

The objective of this study is to evaluate AIIS morphology using ultrasound as compared to golden standard (MRI)

ELIGIBILITY:
Inclusion Criteria:

* adult patients (18 years and older) admitted to the TLVMC sports medicine outpatient clinic due to

hip related complaints

Exclusion Criteria:

* Patient refusal

  * Inability to consent
  * Unavailable 3d imaging the hip joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
AIIS morpholgy | through study completion, an average of 1 year
  AIIS morphology is determined according to the hetzroni classification

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hapa O, Bedi A, Gursan O, Akar MS, Guvencer M, Havitcioglu H, Larson CM. Anatomic footprint of the direct head of the rectus femoris origin: cadaveric study and clinical series of hips after arthroscopic anterior inferior iliac spine/subspine decompression. Arthroscopy. 2013 Dec;29(12):1932-40. doi: 10.1016/j.arthro.2013.08.023. Epub 2013 Oct 18. PMID 24140143
- [Background] Ryan JM, Harris JD, Graham WC, Virk SS, Ellis TJ. Origin of the direct and reflected head of the rectus femoris: an anatomic study. Arthroscopy. 2014 Jul;30(7):796-802. doi: 10.1016/j.arthro.2014.03.003. Epub 2014 May 2. PMID 24793210
- [Background] Lee WA, Saroki AJ, Loken S, Trindade CA, Cram TR, Schindler BR, LaPrade RF, Philippon MJ. Radiographic Identification of Arthroscopically Relevant Acetabular Structures. Am J Sports Med. 2016 Jan;44(1):67-73. doi: 10.1177/0363546515612083. Epub 2015 Nov 20. PMID 26589837